CLINICAL TRIAL: NCT05646940
Title: Fact-based Nutrition for Infants and Lactating Mothers - The NUTRISHIELD Study
Brief Title: Fact-based Nutrition for Infants and Lactating Mothers
Acronym: NUTRISHIELD
Status: Completed | Type: Observational
Sponsor: Instituto de Investigacion Sanitaria La Fe (Other)
Responsible Party: Principal Investigator, Julia Kuligowski, Principal Investigator, Instituto de Investigacion Sanitaria La Fe
Other Study IDs: 818110
Record Dates: First submitted 2022-12-02; First posted 2022-12-12 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Prematurity
Keywords: Prematurity; Nutrition; Preterm infants; Breastfeeding; Human Milk
MeSH Terms: conditions — Premature Birth; Breast Feeding

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Buccal swab, cord blood, human milk, urine, faeces
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- PI-OMM: 25 PI fed with OMM and their mothers
- PI-DHM: 25 PI fed with DHM and their mothers
- TI-OMM: 25 TI fed with OMM and their mothers as control group

SUMMARY:
Human milk (HM) is the ideal source of nutrients for infants, but its composition is highly variable. When not enough own mother's milk (OMM) is available, the administration of pasteurized donor human milk (DHM) is considered the best alternative for feeding preterm infants (PI). The aim of this study is to evaluate the influence of diet, lifestyle habits, psychological stress, and pasteurization on the milk composition, and how it modulates infant's growth, health, and development. NUTRISHIELD is a prospective mother-infant birth cohort in the Spanish-Mediterranean area including three groups: PI <32 weeks of gestation (i) exclusively receiving OMM (i.e., >80% v/v of total intake), and (ii) exclusively receiving DHM, and (iii) term infants (TI) exclusively receiving OMM, as well as their mothers, and HM donors. Biological samples and nutritional, clinical, and anthropometric characteristics are collected at six time points covering the period from birth and until six months of infant's age (complete enteral nutrition (CEN) / recovery birth weight (RBW), and one, two, three, and six months). An additional assessment at two years (corrected age for PI) is conducted, in order to study long-term effects on neurodevelopment.

DETAILED DESCRIPTION:
The genotype, metabolome, and microbiota as well as the HM composition (i.e., macronutrients, fatty acids, vitamins, human milk oligosaccharides, and steroids) are characterized. Portable sensor prototypes for the analysis of HM and urine are benchmarked. Additionally, maternal psychosocial status is measured at the beginning of the study and at month six, including social support, family functioning, perceived stress, anxiety, and depression symptoms, and traumatic life events. Mother-infant postpartum bonding and parental stress is also examined. At six months (corrected age for preterm groups), infant neurodevelopment scales are applied. Mother's concerns and attitudes to breastfeeding are also registered through a specific questionnaire at CEN/RBW and six months. An additional assessment at two years (corrected age for PI) is conducted, in order to study long-term effects on neurodevelopment. Current knowledge on the importance of diet and other environmental factors for infant growth, health, and development is limited and donor-matching at HM banks is frequently only based on gestational age and total protein content of HM. NUTRISHIELD provides an in-depth longitudinal study of the mother-infant-microbiota triad combining multiple biological matrices, newly developed analytical methods, and ad-hoc designed sensor prototypes with a wide range of clinical outcome measures. Data obtained from this study will be used to train a machine-learning algorithm for providing dietary advice to lactating mothers and will be implemented in a user-friendly platform based on a combination of user-provided information and biomarker analysis. A better understanding of the factors affecting the milk's composition, together with the health implications for infants plays an important role in developing improved strategies of nutraceutical management in infant care.

ELIGIBILITY:
Inclusion Criteria:

* Acceptance of the mother to participate and sign an informed consent form
* A gestational age < 32 weeks for the group of PI and > 37 weeks for the group of TI
* Exclusive consumption (i.e., >80% v/v of total intake) of either OMM or DHM.

Exclusion Criteria:

* Non-compliance with any of the inclusion criteria
* The requirement of a special diet for the mother (e.g., celiac disease, diabetes) or maternal consumption of probiotics
* The need of intestinal surgery, severe congenital malformations, or chromosomopathies of the infant
* Mother's residence outside the Valencian Community
* Severe language barriers hampering the collection of necessary data from mothers not speaking Spanish and/or English

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Three mother-infant groups were enrolled, i.e., PI-OMM, PI-DHM, and TI-OMM, and their mothers.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Maternal nutrition and HM composition | From birth to 6 months
  Evaluate associations between the mother's diet and HM composition in PI and TI (i.e., how the potential association between mother's diet and HM nutrient composition is affected by prematurity), and between HM composition and mother's physical and psychosocial status (e.g., lifestyle, perceived stress, anxiety and depression)
HM pasteurization | Up to 6 months
  To evaluate the effect of pasteurization/storage on DHM composition
Infants' health | From birth to month 24
  To evaluate associations between HM composition (OMM or DHM) on growth and other health parameters in PI and TI

CONTACTS AND LOCATIONS:
Overall Officials: Julia Kuligowski, Principal Investigator — Instituto de Investigación Sanitaria La Fe
Locations (1):
- Instituto de Investigación Sanitaria La Fe, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ten-Domenech I, Ramos-Garcia V, Pineiro-Ramos JD, Gormaz M, Parra-Llorca A, Vento M, Kuligowski J, Quintas G. Current Practice in Untargeted Human Milk Metabolomics. Metabolites. 2020 Jan 22;10(2):43. doi: 10.3390/metabo10020043. PMID 31979022
- [Background] Ramos-Garcia V, Ten-Domenech I, Albiach-Delgado A, Gomez-Ferrer M, Sepulveda P, Parra-Llorca A, Campos-Berga L, Moreno-Gimenez A, Quintas G, Kuligowski J. Isolation and Lipidomic Screening of Human Milk Extracellular Vesicles. Methods Mol Biol. 2023;2571:177-188. doi: 10.1007/978-1-0716-2699-3_18. PMID 36152162
- [Background] Ten-Domenech I, Ramos-Garcia V, Moreno-Torres M, Parra-Llorca A, Gormaz M, Vento M, Kuligowski J, Quintas G. The effect of Holder pasteurization on the lipid and metabolite composition of human milk. Food Chem. 2022 Aug 1;384:132581. doi: 10.1016/j.foodchem.2022.132581. Epub 2022 Feb 26. PMID 35257998
- [Background] Pineiro-Ramos JD, Parra-Llorca A, Ten-Domenech I, Gormaz M, Ramon-Beltran A, Cernada M, Quintas G, Collado MC, Kuligowski J, Vento M. Effect of donor human milk on host-gut microbiota and metabolic interactions in preterm infants. Clin Nutr. 2021 Mar;40(3):1296-1309. doi: 10.1016/j.clnu.2020.08.013. Epub 2020 Aug 19. PMID 32863061
- [Background] Poulimeneas D, Bathrellou E, Antonogeorgos G, Mamalaki E, Kouvari M, Kuligowski J, Gormaz M, Panagiotakos DB, Yannakoulia M; NUTRISHIELD Consortium. Feeding the preterm infant: an overview of the evidence. Int J Food Sci Nutr. 2021 Feb;72(1):4-13. doi: 10.1080/09637486.2020.1754352. Epub 2020 Apr 27. PMID 32340495
- [Background] Ramos-Garcia V, Ten-Domenech I, Vento M, Bullich-Vilarrubias C, Romani-Perez M, Sanz Y, Nobili A, Falcone M, Di Stefano M, Quintas G, Kuligowski J. Fast profiling of primary, secondary, conjugated, and sulfated bile acids in human urine and murine feces samples. Anal Bioanal Chem. 2023 Aug;415(20):4961-4971. doi: 10.1007/s00216-023-04802-8. Epub 2023 Jun 20. PMID 37338567
- [Result] Ramos-Garcia V, Ten-Domenech I, Moreno-Gimenez A, Campos-Berga L, Parra-Llorca A, Solaz-Garcia A, Lara-Canton I, Pinilla-Gonzalez A, Gormaz M, Vento M, Kuligowski J, Quintas G. GC-MS analysis of short chain fatty acids and branched chain amino acids in urine and faeces samples from newborns and lactating mothers. Clin Chim Acta. 2022 Jul 1;532:172-180. doi: 10.1016/j.cca.2022.05.005. Epub 2022 May 8. PMID 35545167
- [Result] Akhgar CK, Nurnberger V, Nadvornik M, Ramos-Garcia V, Ten-Domenech I, Kuligowski J, Schwaighofer A, Rosenberg E, Lendl B. Fatty Acid Determination in Human Milk Using Attenuated Total Reflection Infrared Spectroscopy and Solvent-Free Lipid Separation. Appl Spectrosc. 2022 Jun;76(6):730-736. doi: 10.1177/00037028211065502. Epub 2022 Feb 4. PMID 35119320
- [Result] Ramos-Garcia V, Ten-Domenech I, Moreno-Gimenez A, Campos-Berga L, Parra-Llorca A, Ramon-Beltran A, Vaya MJ, Mohareb F, Molitor C, Refinetti P, Silva A, Rodrigues LA, Rezzi S, Hodgson ACC, Canarelli S, Bathrellou E, Mamalaki E, Karipidou M, Poulimeneas D, Yannakoulia M, Akhgar CK, Schwaighofer A, Lendl B, Karrer J, Migliorelli D, Generelli S, Gormaz M, Vasileiadis M, Kuligowski J, Vento M. Fact-based nutrition for infants and lactating mothers-The NUTRISHIELD study. Front Pediatr. 2023 Apr 18;11:1130179. doi: 10.3389/fped.2023.1130179. eCollection 2023. PMID 37144153
- [Result] Ramos-Garcia V, Ten-Domenech I, Moreno-Gimenez A, Campos-Berga L, Parra-Llorca A, Gormaz M, Vento M, Karipidou M, Poulimeneas D, Mamalaki E, Bathrellou E, Kuligowski J. Joint Microbiota Activity and Dietary Assessment through Urinary Biomarkers by LC-MS/MS. Nutrients. 2023 Apr 14;15(8):1894. doi: 10.3390/nu15081894. PMID 37111113